CLINICAL TRIAL: NCT04791293
Title: Predictive Value of MELD-Na Score for Perioperative Complications in Non-cirrhotic Patients With Gastric Cancer
Brief Title: The Model for End-Stage Liver Disease Sodium (MELD-Na) Score in Non-cirrhotic Patients With Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cihad Tatar, Associate Professor, Istanbul Training and Research Hospital
Other Study IDs: 2630
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer; Complication,Postoperative; Complications; Gastrointestinal, Postoperative; Morality
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with postoperative complications
  Interventions: Other: MELD-Na score
- Group 2: Patients without postoperative complications
  Interventions: Other: MELD-Na score

INTERVENTIONS:
Other: MELD-Na score — MELD-Na scores will be compared between the groups

SUMMARY:
Gastric cancer is the fifth most common cancer worldwide. Gastrectomy with lymphadenectomy is still the most effective treatment modality, depending on the stage and location. Despite many radiological, surgical and anesthetic innovations, serious complications such as anastomotic leakage, intra-abdominal abscesses, wound complications are seen secondary to gastrectomy. Many clinical studies have been conducted to prevent and predict these complications.

The Model for End-Stage Liver Disease (MELD) score, in which bilirubin, international normalized ratio (INR) and serum creatinine values were used to determine surgical risks in patients scheduled for liver transplantation. Latter developed by adding serum sodium (Na) to the formula. The MELD-Na score is used to predict postoperative complications in non-cirrhotic patients because of its simple and easy calculation.Moreover, The Meld-Na score was later used to predict complications for surgical procedures other than liver surgery such as colorectal surgery.

In this study, we aimed to investigate the importance of the Meld-Na score in predicting the perioperative and postoperative outcomes in patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastrectomy due to gastric cancer

Exclusion Criteria:

* Patients with pulmonary, hepatic and renal disfunctions,
* Patients with diagnosed with a different cancer in the last 5 years and
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing gastrectomy due to gastric cancer
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
MELD-Na score difference between the groups | 30 days
  Importance of MELD-Na score in predicting postoperative complications in patients with gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Cihad Tatar, MD, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coakley KM, Sarasani S, Prasad T, Steele SR, Paquette I, Heniford BT, Davis BR. MELD-Na Score as a Predictor of Anastomotic Leak in Elective Colorectal Surgery. J Surg Res. 2018 Dec;232:43-48. doi: 10.1016/j.jss.2018.04.012. Epub 2018 Jul 2. PMID 30463752
- [Background] Schlosser KA, Kao AM, Zhang Y, Prasad T, Kasten KR, Davis BR, Heniford BT, Colavita PD. MELD-Na score associated with postoperative complications in hernia repair in non-cirrhotic patients. Hernia. 2019 Feb;23(1):51-59. doi: 10.1007/s10029-018-1849-2. Epub 2018 Nov 16. PMID 30446849
- [Background] Yasri S, Wiwanitkit V. MELD-Na score and postoperative complications in hernia repair. Hernia. 2019 Aug;23(4):823. doi: 10.1007/s10029-019-01886-z. Epub 2019 Jan 22. No abstract available. PMID 30671898